CLINICAL TRIAL: NCT02836106
Title: Postprandial Effects of High-fat Meals With Different Dairy Products on Lipid Metabolism and Inflammation in Healthy and Obese Subjects
Brief Title: Postprandial Effects of High-fat Meals With Different Dairy Products on Lipid Metabolism and Inflammation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oslo (Other)
Collaborators: Tine (Industry); The Research Council of Norway (Other)
Responsible Party: Principal Investigator, Stine Marie Ulven, Professor, University of Oslo
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: 2016/418/REK sør-øst B
Record Dates: First submitted 2016-06-08; First posted 2016-07-18 (Estimated); Last update posted 2022-11-07 (Actual); Status verified 2022-11

CONDITIONS: Healthy; Overweight; Obesity
Keywords: Healthy Volunteers; Obese Volunteers
MeSH Terms: conditions — Overweight; Obesity | interventions — Butter; Cheese

ARMS (2):
- Healthy (Experimental): Lean subjects (BMI<25) with a waist circumference of <94 cm for men and<80 cm for women. Subjects will be randomly assigned to eat butter, cheese, whipped cream and sour cream in a cross-over design.
  Interventions: Other: Butter; Other: Cheese; Other: Whipped cream; Other: Sour cream
- Obese (Experimental): Overweight and obese subjects (BMI≥25) with a waist circumference of ≥94 cm for men and ≥80 cm for women. Subjects will be randomly assigned to eat butter, cheese, whipped cream and sour cream in a cross-over design.
  Interventions: Other: Butter; Other: Cheese; Other: Whipped cream; Other: Sour cream

INTERVENTIONS:
Other: Butter — Butter with jam and three slices of bread
Other: Cheese — Cheese with jam and three slices of bread
Other: Whipped cream — Whipped cream with jam and three slices of bread
Other: Sour cream — Sour cream with jam and three slices of bread

SUMMARY:
The aim of this project is to elucidate how high-fat meals with different kinds of dairy products affect postprandial responses of lipid metabolism and inflammatory markers in healthy and obese subjects.

ELIGIBILITY:
Inclusion Criteria:

* The study will include both men and women aged 18-70 years with the aim of an even age and gender balance.
* Participants in the healthy group will need to have a body mass index (BMI) between 18.5 - 24.9 kg/m2 and a waist circumference (WC) of <94 cm for men and<80 cm for women.
* Participants in the obese group will need to have a BMI of ≥25 kg/m2 and a waist circumference of ≥94 cm for men and ≥80 cm for women.
* All subjects must be willing to eat three slices of bread with a dairy product and jam as breakfast.

Exclusion Criteria:

* BMI <18.5 kg/m2 or >25 kg/m2 in the healthy group and <25 kg/m2 in the obese group
* WC ≥94 for men and ≥80 cm for women in the healthy group, <94/80 cm for men/women in the obese group
* Weight change of ± 5 % of body weight in the last three months
* TG ≥1.3 mmol/L in the healthy group
* CRP >10 mg/L
* Total cholesterol >6.1 mmol/L for subjects 18-29 years, >6.9 mmol/L for subjects 30-49 years and >7.8 mmol/L for subjects ≥50 years old
* Blood pressure >160/100 mm Hg
* Comorbidities including diabetes type I and II (blood glucose ≥7 mmol/L fasting), coronary heart disease, haemophilia, anaemia (hemoglobin <120 gram/L), gastro intestinal disease and hyperthyroidism (TSH >4 mU/L)
* Pregnant or lactating
* Allergic or intolerant to gluten, milk protein and/or lactose
* Use of medications affecting lipid metabolism or inflammation
* Unwilling to seponate omega-3 rich supplements four weeks prior to screening and during the study period
* Hormone treatment (stabile dose of contraception or thyroxin for the last three months excepted)
* Blood donation two months prior to test day 1 or during the study period
* Tobacco smoking
* Excessive regular alcohol consumption (>40 grams per day) or prior to the test day

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2016-06; Primary Completion 2017-04 (Actual); Study Completion 2017-04 (Actual)

PRIMARY OUTCOMES:
Changes in levels of circulating triglycerides | Measured at baseline and 2,4 and 6 hours after intake of test meal

SECONDARY OUTCOMES:
Changes in total cholesterol and lipoproteins | Measured at baseline and 2,4 and 6 hours after intake of test meal
  Changes in total cholesterol and lipoproteins, such as low-density lipoprotein and high-density lipoprotein
Changes in levels of apolipoproteins | Measured at baseline and 2,4 and 6 hours after intake of test meal
  Changes in levels of apolipoproteins, i.e. apo A1, apo B, apo B-48 and apo C-III
Changes in levels of free fatty acids | Measured at baseline and 2,4 and 6 hours after intake of test meal
Changes in levels of circulating inflammatory markers | Measured at baseline and 2,4 and 6 hours after intake of test meal
  Changes in levels of inflammatory markers, such as cytokines, acute phase proteins and soluble adhesion molecules
Changes in levels of circulating endotoxins | Measured at baseline and 2,4 and 6 hours after intake of test meal
Changes in gene expressions (mRNA and microRNA) of genes related to lipid metabolism and inflammation in Peripheral Blood Mononuclear Cells (PBMC) | Measured at baseline and 2,4 and 6 hours after intake of test meal
Changes in whole genome transcriptomics in PBMC | Measured at baseline and 2,4 and 6 hours after intake of test meal
Check DNA for Single Nucleotide Polymorphisms related to responses of a high-fat meal | Measured at baseline and 2,4 and 6 hours after intake of test meal
Examine epigenetics through DNA methylation and histone modification | Measured at baseline and 6 hours after intake of test meal
Changes of plasma and urine metabolomics | Measured at baseline and 2,4 and 6 hours after intake of test meal
  Changes in levels of metabolites, such as glucose and amino acids
Changes in levels of gut hormones | Measured at baseline and 2,4 and 6 hours after intake of test meal
  Changes in levels of gut hormones, such as peptide YY (PYY)
Changes in experiences of hunger and satiety by Visual Analogue Scales (VAS) questionnaire | Measured at baseline and 2,4 and 6 hours after intake of test meal

CONTACTS AND LOCATIONS:
Overall Officials: Stine M Ulven, PhD, Principal Investigator — University of Oslo
Locations (1):
- University of Oslo, Oslo, Norway

REFERENCES:
- [Derived] Hansson P, Holven KB, Oyri LKL, Brekke HK, Gjevestad GO, Thoresen M, Ulven SM. Sex differences in postprandial responses to different dairy products on lipoprotein subclasses: a randomised controlled cross-over trial. Br J Nutr. 2019 Oct 14;122(7):780-789. doi: 10.1017/S0007114519001429. PMID 31208475
- [Derived] Hansson P, Holven KB, Oyri LKL, Brekke HK, Biong AS, Gjevestad GO, Raza GS, Herzig KH, Thoresen M, Ulven SM. Meals with Similar Fat Content from Different Dairy Products Induce Different Postprandial Triglyceride Responses in Healthy Adults: A Randomized Controlled Cross-Over Trial. J Nutr. 2019 Mar 1;149(3):422-431. doi: 10.1093/jn/nxy291. PMID 30759235